CLINICAL TRIAL: NCT05566678
Title: A 12-month, 3-group, Preference, Multi-center Study to Demonstrate the Effects of Switching From Cigarettes to Tobacco Heating System (THS) on Systemic Endothelial Function in Subjects With Established Atherosclerotic Disease
Brief Title: Effect of Switching From Cigarette Smoking to THS on Systemic Endothelial Function in Subjects With Established Atherosclerotic Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped before enrollment, after a feasibility review revealed we would be unable to measure the primary endpoint (flow mediated dilation - FMD) with a high degree of reproducibility and minimum variability in a multi-country setting.
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P1-CVD-05
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases; Smoking; Tobacco Use; Peripheral Arterial Disease; Coronary Artery Disease
Keywords: Flow Mediated Dilation; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Smoking; Tobacco Use; Peripheral Arterial Disease; Coronary Artery Disease; Atherosclerosis | interventions — Tobacco Products

STUDY DESIGN:
Intervention Model Description: A three-group ambulatory preference design, multi-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cigarette (Active Comparator): Smokers who self-selected to continue smoking cigarettes.
  Interventions: Other: Cigarette
- Tobacco Heating System (Active Comparator): Smokers who self-selected to switch to THS use.
  Interventions: Other: THS
- Smoking Abstinence (Active Comparator): Smokers who self-selected to abstain from smoking.
  Interventions: Other: Smoking Abstinence

INTERVENTIONS:
Other: Cigarette — Subjects who self-selected to continue smoking their own preferred brand of commercially available cigarettes.
  Arms: Cigarette
Other: THS — Subjects who self-selected to quit smoking during the study duration will switch from cigarettes to using THS.
  Other Names: Tobacco Heating System 3.0
  Arms: Tobacco Heating System
Other: Smoking Abstinence — Subjects who self-selected to quit smoking may be prescribed Nicotine Replacement Therapy (NRT) to support them in remaining abstinent from use of any tobacco and nicotine containing products during the study. (Behavioral support will be provided to subjects to aid with abstinence.)
  Arms: Smoking Abstinence

SUMMARY:
The purpose of this study is to demonstrate improvement in flow mediated dilation (FMD), a functional endpoint associated with the progression of atherosclerosis, when switching from cigarettes to the Tobacco Heating System (THS) in subjects with peripheral arterial disease (PAD) and/or coronary artery disease (CAD). The study is planned to be conducted in the US, Europe, and Asia.

DETAILED DESCRIPTION:
The goal of this longitudinal study is to demonstrate improvement in FMD, a functional endpoint associated with the progression of atherosclerosis and a predictor of future cardiovascular (CV) events in subjects with PAD and/or CAD, when switching from cigarettes to THS. Other CV functional endpoints, or cardiovascular biomarkers of potential harm (BoPH) representative of different pathophysiologic pathways associated with increased CV risk in smokers with established atherosclerosis will be assessed. It is expected that the totality of the evidence from this study will show the potential of THS to slow down the progression of atherosclerosis, thus helping to delay a CV event, or delaying a secondary event.

ELIGIBILITY:
Main Inclusion Criteria:

* History of coronary artery disease, defined as documented CAD (stable) with coronary artery stenosis on coronary angiogram ≥50% (incl. Percutaneous Coronary Intervention (PCI) / Coronary artery bypass graft surgery (CABG)) in the medical history or previously documented acute coronary syndrome (ACS) / myocardial infarction occurring more than 1 month prior to V1. AND / OR, History of peripheral artery disease (PAD) defined as ABI <0.9 or TBI <0.6 or clinical diagnosis of chronic, symptomatic lower limb ischemia as defined by Fontaine's stages I, IIa and IIb.
* Body mass index (BMI) 17.6-40.0 kg/m2 and body weight > 50 kg (male) or 40 kg (female).
* Subject has a smoking history of at least 10 years.
* Subject has not used other tobacco and nicotine products apart from cigarettes on a daily basis over the past year prior to V1.
* Subject has been smoking ≥ 10 commercially available cigarettes/day on average (no brand restriction) for at least 1 year prior to V1 (based on self-reporting).
* For subjects not willing to quit smoking only: have been advised to quit smoking and informed of smoking risks and of cessation programs and is still not willing to quit during the study duration.
* Subjects willing to quit smoking only: willing to and set a target quit date (TQD) within the next 28 days at V1 as assessed by self-reported questions

Main Exclusion Criteria:

* Planned peripheral or coronary intervention or surgical procedure.
* Unstable angina pectoris.
* Critical limb ischemia (absolute peripheral pressures <50mmHg).
* Recent (< 30 days) PAD revascularization therapy prior to V1.
* Recent ACS / myocardial infarction or stroke / TIA <30 days prior to V1.
* Pre-existing symptomatic heart failure with reduced ejection fraction (EF<35%).
* Planned peripheral or coronary intervention or surgical procedure related to CAD or PAD.
* Subjects with spirometry values indicating chronic obstructive pulmonary disease (COPD) GOLD* Stage 3 or 4 (FEV1/FVC <0.7 & FEV1 <50% predicted [post-BD])
* Existing known serious infection or chronic inflammatory systemic disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, uncontrolled diabetes (HbA1c ≥ 7.0 % [or ≥ 53.0 mmol/mol]) or uncontrolled hypertension (systolic blood pressure≥140 mmHg and / or diastolic blood pressure ≥90 mmHg., stage 4 and 5 chronic kidney disease, etc…).
* Currently active cancer or history of cancer within the last 5 years prior to V1.
* History of alcohol and / or drug abuse (other than tetrahydrocannabinol [THC]).
* Positive serology test (human immunodeficiency virus (HIV) 1/2), hepatitis B and / or C).
* Female subject is pregnant or breastfeeding, (a urine pregnancy test will be performed at V1 and V2)
* Previous participation in this study, or participation in an investigational study (drug or medical device) within 4 weeks before V1 (participation in observational studies/registries allowed)
* For women of childbearing potential, female subject who does not agree to using an acceptable method of effective contraception during the entire study.

[*Global Initiative for Obstructive Lung Disease]

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation | From baseline to 12 months.
  Change from baseline in flow mediated dilation (%FMD) of the brachial artery at 12 months before administration of a vasodilator (nitroglycerin)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.

IPD SHARING:
Plan to Share IPD: No